CLINICAL TRIAL: NCT02435238
Title: AWARE: A World-wide Antihistamine-Refractory Chronic Urticaria Patient Evaluation
Brief Title: AWARE - Chronic Urticaria
Acronym: AWARE
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025EGB01
Record Dates: First submitted 2014-12-02; First posted 2015-05-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non interventional study collecting patient reported outcomes. The study aims to assess the disease burden of chronic urticaria patients and to record the therapies used in daily clinical practice in the UK and the impact they have on the quality of life and work productivity of individual patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be 18 years old Subject must be willing and able to provide written informed consent for collection and analysis of routine data and PROs Subject must have medically confirmed diagnosis of chronic urticaria present for more than 2 months.

Subject must be refactory to at least one H1 antihistamine

Exclusion Criteria:

Subjects who in the estimation of the treating physician are unlikely to be available for the full duration of the follow-up period of 24 months.

Subjects taking must not take part in any other concurrent urticarial study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Urticaria Patients
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Measuring responses to PROs from patients on different treatments | 24 months
  Measuring quality of life, work productivity and changes in disease for patients on different treatment.

SECONDARY OUTCOMES:
To record use of clinical resources | 24 months
  Measuring how often clinical resources (hospitalisations, frequency of visits) are used
Previous, current and future medication | 24 months
  Recording medication use throughout the 24 months
The disease burden of chronic urticaria | 24 months
  The "disease burden" (including impact on sleep and work productivity)
Rates of spontaneous remission | 24 months
Treatment algorithms and trends | 24 months
  Measuring treatment algorithms and trends during the study course (including therapy adjustments and duration of use of each substance class)
Co-morbidities of refractory CU patients | 24 months
first onset of chronic urticaria | 24 months
  Time of first onset of the disease and number physicians consulted
Number of patients with angiodema | 24 months
Number of angioedema episodes during the observational phase | 24 months
Prevalence of inducible urticaria | 24 months
  The number of patients in the study population that are diagnosed with inducible urticaria.
Diagnosis of CSU | 24 months

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Darlington, Durham
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Coventry, Warwickshire
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chester
  - Novartis Investigative Site, Durham
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Sheffield